CLINICAL TRIAL: NCT01837706
Title: The Impact of Emergency Physician Empathy on Litigation Propensity
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Dustin Smith, Faculty, Loma Linda University
Other Study IDs: RS-5120206
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Empathy
Keywords: Empathy; Communication; Physician litigation
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Emergency Room Patients

SUMMARY:
The purpose of this study is to observe whether people would report being less likely to sue a physician who shows more empathy when giving a patient potentially bad news regarding their medical condition.

DETAILED DESCRIPTION:
The investigators hypothesized that patients will have less propensity to sue emergency physicians after a poor outcome if the physician demonstrated empathy by verbalizing that they recognize the patient is concerned about their symptoms, and that the patient knows their typical state of health better than a physician seeing them for the first time. Accordingly, the investigators will assess whether the presence or absence of emergency physician empathetic statements in videotaped simulated encounters will alter patient propensity towards litigation. Secondary objectives are to assess whether the presence or absence of empathetic statements alters patient perceptions of discharge instruction clarity, physician expertness, physician caring, and physician desirability.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Room Patient

Exclusion Criteria:

* Non-English speaking
* Not healthy enough to be in waiting room

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Emergency room patients
Sampling Method: Probability Sample
Enrollment: 437 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Intention to sue | Immediately after viewing
  This outcome will be assessed by asking "Would you sue this doctor?" after viewing a short video. Items will be measured on a 5-point scale (1=Definitely no to 5=Definitely yes).

SECONDARY OUTCOMES:
Assessment of physician expertise | Immediately after viewing
  This outcome will be assessed by asking "Do you believe this physician is an expert?" after viewing a short video. Items will be measured on a 5-point scale (1=Definitely no to 5=Definitely yes).
Assessment of physician caring | Immediately after viewing
  This outcome will be assessed by asking "Do you think this doctor cared about the patient?" after viewing a short video. Items will be measured on a 5-point scale (1=Definitely no to 5=Definitely yes).
Assessment of whether subject would want to be physician's patient | Immediately after viewing
  This outcome will be assessed by asking "Would you want this physician as your doctor?" after viewing a short video. Items will be measured on a 5-point scale (1=Definitely no to 5=Definitely yes).
Assessment of clarity of physician instructions | Immediatley after viewing
  This outcome will be assessed by asking "Did you understand the instructions the doctor gave the patient?" after viewing a short video. Items will be measured on a 5-point scale (1=Definitely no to 5=Definitely yes).

CONTACTS AND LOCATIONS:
Overall Officials: Dustin Smith, MD, Principal Investigator — Loma Linda University; Ellen Reibling, PhD, Study Director — Loma Linda University; Jesse Kellar, MD, Study Director — Loma Linda University; Steve Green, MD, Study Director — Loma Linda University; Elizabeth Walters, MD, Study Director — Loma Linda University
Locations (1):
- Loma Linda University Emergency Department, Loma Linda, California, United States

REFERENCES:
- [Derived] Smith DD, Kellar J, Walters EL, Reibling ET, Phan T, Green SM. Does emergency physician empathy reduce thoughts of litigation? A randomised trial. Emerg Med J. 2016 Aug;33(8):548-52. doi: 10.1136/emermed-2015-205312. Epub 2016 Mar 21. PMID 27002161